CLINICAL TRIAL: NCT03415464
Title: Prevention of Musculoskeletal Injuries in Slovenian Armed Forces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Vedran Hadzic, Head of the Sports Medicine Department, Faculty of Sport, University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 630-1/2016-3
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Knee Injuries and Disorders; Ankle Injuries and Disorders; Low Back Pain
MeSH Terms: conditions — Knee Injuries; Disease; Ankle Injuries; Low Back Pain | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional training (Experimental): 15 weeks of structured exercise intervention in the form of functional training. We have divided 15 weeks into 5 cycles each cycle lasting 3 weeks. Intervention will be administered twice per week, and each session will last 45 minutes.Each 45 minutes will be further divided into 10 minutes of functional warm-up, 30 minutes of neuromuscular training (strength, agility, balance, coordination) and 5 minutes of cool down. During the 3 week period the intensity of exercise will be increased with different form of same exercise, different number of repetitions and exercise duration.
  Interventions: Other: Exercise
- Regular army training (No Intervention): Regular military training.

INTERVENTIONS:
Other: Exercise — neuromuscular training
  Arms: Functional training

SUMMARY:
Physical readiness of military personnel is a cornerstone of any army, as soldiers are expected to meet high physical demands on a daily basis, and soldiers must complete one hour of physical conditioning each day. Participation in physical conditioning increases the risk of musculoskeletal injuries, and our 10-year retrospective analysis shows that 5% of soldiers sustain a sports injury during physical conditioning each year, and that ankle and knee injuries have the highest incidence rates of 25% and 20%, respectively. The primary objective of our study is to decrease the rate of ankle and knee injuries by implementing a preventive training program. The study is designed as a prospective randomized controlled trial with two arms (experimental and control).

DETAILED DESCRIPTION:
Members of Slovenian Armed Forces - SAF (age range 18-51 years) are expected to participate in the study. Prior to recruitment the whole project will be explained to soldiers in a form of briefing during which they have the opportunity to ask and have answers to any questions concerning the nature of subsequent research. Following that explanation each participant will sign a consent form to voluntarily participate. No compensation will be given or promised for participation in a study that was approved by the Ethical board of the Faculty of Sport in Ljubljana (No. 454/2017). At the time of testing all soldiers must be free of acute injuries and should not reported any pain in musculo-skeletal system. Prior to the implementation of the preventive program all participants will underwent the set of functional testing that includes counterMovement jump (CMJ) testing, stork balANce test, pUll-ups, single leg hAmstrings bridge test, and loaded prone pLank test - MANUAL. Following initial testing a 15-week preventive training program will be implemented in experimental group, while control group will be training as usual. Following the intervention final testing will be performed to check for effectiveness of the intervention. After that a follow-up period will start during which injuries will be registered in both groups and later compared between groups (control and experimental) and within (2016-2017 injuries) groups to see if incidence rate of ankle and knee injuries has fallen.

ELIGIBILITY:
Inclusion Criteria:

* no major injuries that would require more than 4 weeks to recover upon entry into the study
* age >18 y
* finished initial Army training

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University in Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Background] Kovcan B, Vodicar J, Simenko J, Videmsek M, Pori P, Vedran H. Retrospective and Cross-sectional Analysis of Physical Training-Related Musculoskeletal Injuries in Slovenian Armed Forces. Mil Med. 2019 Jan 1;184(1-2):e195-e199. doi: 10.1093/milmed/usy156. No abstract available. PMID 29982738
- [Result] Vodicar M, Kovcan B, Pori P, Vodicar J, Simenko J, Karpljuk D, Markovic G, Hadzic V. Regular strength training and baseline fitness in overweight infantry members of Slovenian Armed Forces. BMJ Mil Health. 2022 Apr;168(2):141-145. doi: 10.1136/bmjmilitary-2020-001451. Epub 2020 Jun 2. PMID 32487675
- [Result] Simenko J, Kovcan B, Pori P, Vodicar J, Vodicar M, Hadzic V. The Relationship Between Army Physical Fitness and Functional Capacities in Infantry Members of the Slovenian Armed Forces. J Strength Cond Res. 2021 Dec 1;35(12):3506-3512. doi: 10.1519/JSC.0000000000003344. PMID 31800475
- [Result] Kozinc Z, Sarabon N, Kovcan B, Simenko J, Pori P, Vodicar J, Hadzic V. Effects of 12-week full body resistance exercise on vertical jumping with and without military equipment in Slovenian Armed Forces. BMJ Mil Health. 2023 Oct;169(5):391-396. doi: 10.1136/bmjmilitary-2021-001899. Epub 2021 Sep 7. PMID 34493610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from January to February 2017.
Pre-assignment Details: Initially, there were 160 soldier who approved to participate in initial testing, but prior to assignment of participants to groups 55 of them has declined further participation for different reasons, so only 105 soldiers was later randomised into groups, but the completion rate after this point was 100%.
Period: Overall Study
Arm/Group | Functional Training | Regular Army Training
Started | 64 | 41
Completed | 64 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Functional Training: 15 weeks of structured exercise intervention in the form of functional training. We have divided 15 weeks into 5 cycles each cycle lasting 3 weeks. Intervention was administered twice per week, and each session lasted 45 minutes. Each 45 minutes was further divided into 10 minutes of functional warm-up, 30 minutes of neuromuscular training (strength, agility, balance, coordination) and 5 minutes of cool down. During the 3 week period the intensity of exercise was increased with different form of same exercise, different number of repetitions and exercise duration.
  Exercise: neuromuscular training
- Total: Total of all reporting groups
Arm/Group | Functional Training | Regular Army Training | Total
Number analyzed (Participants) | 64 | 41 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6) | 34 (6) | 32 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 63 | 37 | 100
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 41 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Single leg bridge test (right leg) [Mean (Standard Deviation); unit: number of repetitions] | 26 (9) | 27 (7) | 27 (8)
Single leg bridge test (left leg) [Mean (Standard Deviation); unit: number of repetitions] | 25 (8) | 25 (7) | 25 (8)
Loaded prone plank [Mean (Standard Deviation); unit: time in seconds] | 119 (48) | 115 (50) | 117 (49)
Pull ups [Mean (Standard Deviation); unit: number of repetitions] | 4 (4) | 4 (4) | 4 (4)
Stork balance test (right leg) [Mean (Standard Deviation); unit: time in seconds] | 14 (13) | 13 (14) | 14 (13)
Stork balance test (left leg) [Mean (Standard Deviation); unit: time seconds] | 14 (13) | 13 (13) | 14 (13)
Countermovement jump height [Mean (Standard Deviation); unit: centimeters] | 28.3 (3.9) | 26.0 (4.9) | 27.4 (4.5)
Loaded countermovement jump height [Mean (Standard Deviation); unit: centimeters] | 25.2 (3.3) | 23.5 (5.1) | 24.6 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Soldiers With Ankle and Knee Injuries
Description: Percentage of soldiers with ankle and knee injuries during the study period.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Functional Training | Regular Army Training
Number analyzed (Participants) | 64 | 41
Participants | 1 | 3
Statistical Analysis 1: Comparison: Functional Training vs Regular Army Training; Test type: Other; p = 0.134, Chi-squared

2. Secondary Outcome: Vertical Jump Performance
Description: jump height in countermovement jump
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Functional Training | Regular Army Training
Number analyzed (Participants) | 64 | 41
centimeters | 35.4 (10.3) | 29.9 (10.8)

3. Secondary Outcome: Pull-ups Performance
Description: number of overhand pull-ups in one minute
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Functional Training | Regular Army Training
Number analyzed (Participants) | 64 | 41
repetitions | 6 (4) | 4 (4)

4. Secondary Outcome: Hamstring Repetitive Strength
Description: Number of single leg raises on the 60 cm box
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: repeitions
Arm/Group | Functional Training | Regular Army Training
Number analyzed (Participants) | 64 | 41
repeitions | 25 (8) | 25 (7)

ADVERSE EVENTS:
Time Frame: 1 year
Description: We were following the possible injury occurrence due to intervention itself. We have not registered any injury to be caused by intervention per se.
Groups:
- Regular Military Training: Regular military training.
Arm/Group | Functional Training | Regular Military Training
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/41
Other Adverse Events (participants affected / at risk) | 0/64 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03415464/Prot_SAP_000.pdf